CLINICAL TRIAL: NCT04075227
Title: A Randomized Clinical Trial: Comparison of the Efficacy of Topical 0.2% Loteprednol Etabonate and Topical 0.1% Dexamethasone in Impending Recurrent Pterygium
Brief Title: Topical 0.2% Loteprednol Etabonate vs. Topical 0.1% Dexamethasone in Impending Recurrent Pterygium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wannisa Suphachearabhan (Other)
Collaborators: Srinakharinwirot University (Other)
Responsible Party: Sponsor-Investigator, Wannisa Suphachearabhan, Principal investigator, Srinakharinwirot University
Organization: Srinakharinwirot University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC006/60
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Pterygium of Eye; Steroid-Induced Glaucoma
Keywords: Impending recurrent pterygium; 0.2% loteprednol etabonate; 0.1% dexamethasone
MeSH Terms: conditions — Pterygium | interventions — Loteprednol Etabonate; Dexamethasone

STUDY DESIGN:
Intervention Model Description: The participants were randomized into 2 groups. Group 1 were treated with subconjunctival 5-FU injection and topical 0.2% loteprednol etabonate while group 2 were treated with subconjunctival 5-FU injection and topical 0.1% dexamethasone (CD-oph: dexamethasone sodium phosphate 1 mg/mL, chloramphenicol 5 mg/mL, tetrahydrozaline hydrochloride 0.25 mg/mL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.2% loteprednol etabonate (Experimental): This group was treated with subconjunctival 5-FU injection and topical 0.2% loteprednol etabonate every 4-6 hours for 4 weeks. After that, the regimen was gradually decreased until cessation at 3 months.
  Interventions: Drug: 0.2% loteprednol etabonate
- 0.1% dexamethasone (Active Comparator): This group was treated with subconjunctival 5-FU injection and topical 0.1% dexamethasone (CD-oph) every 4-6 hours for 4 weeks. After that, the regimen was gradually decreased until cessation at 3 months.
  Interventions: Drug: 0.1% dexamethasone

INTERVENTIONS:
Drug: 0.2% loteprednol etabonate — Use topical 0.2% loteprednol etabonate eyedrop every 4-6 hours for 4 weeks. After that, the regimen was gradually decreased until cessation at 3 months.
  Other Names: Alrex
  Arms: 0.2% loteprednol etabonate
Drug: 0.1% dexamethasone — Use topical 0.1% dexamethasone eyedrop every 4-6 hours for 4 weeks. After that, the regimen was gradually decreased until cessation at 3 months.
  Other Names: CD-oph
  Arms: 0.1% dexamethasone

SUMMARY:
The objective of this study was to evaluate the efficacy of topical 0.2% loteprednol etabonate, a 'soft steroid', compared with topical 0.1% dexamethasone, which is widely used in postoperative pterygium excision to prevent the recurrence of pterygium. If 0.2% loteprednol etabonate is non-inferior in efficacy compared with 0.1% dexamethasone, it may be used postoperatively in pterygium excision patients with the benefit of a low incidence of ocular hypertension or secondary glaucoma.

DETAILED DESCRIPTION:
A prospective randomized control trial was performed from October 2015 to April 2019 at the Department of Ophthalmology, Thammasat Hospital, Thailand and Panyananthaphikkhu Chonprathan Medical Center, Thailand.

Subjects Patients who had pterygium excision with amniotic membrane transplantation (AMT) and who had impending recurrent pterygium stage 3 defined as fibrovascular tissue not invading the cornea were included.

Then the participants were randomized into 2 groups. Both groups received subconjunctival 5-fluorouracil (5-FU) injection 5mg/0.1 mL with 27-gauge needle in the area of fibrovascular tissue, and then the eyes were irrigated with 30 mL of normal saline. 0.2% loteprednol etabonate was prescribed in group 1, and 0.1% dexamethasone (CD-oph) was prescribed in group 2 every 4-6 hours for 4 weeks. After that, the regimen was gradually decreased until cessation at 3 months. 5-FU was repeatedly injected monthly in the presence of marked inflammation and not more than 3 times to prevent complications.

All patients were followed-up at 1, 3, 6, and 9 months to assess the impending recurrent pterygium severity score, intraocular pressure, complications, detection of true recurrent pterygium, and time to recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had pterygium excision with amniotic membrane transplantation and who had impending recurrent pterygium stage 3 defined as fibrovascular tissue not invading the cornea

Exclusion Criteria:

* recurrent pterygium
* received adjunctive treatment with beta radiation, mitomycin C or 5-fluorouracil
* glaucoma or intraocular pressure > 21 mmHg
* history of 5-fluorouracil or chloramphenicol allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
rate of true recurrent pterygium | 6 months
  true recurrent pterygium is the fibrovascular tissue that invade into cornea

SECONDARY OUTCOMES:
severity score of impending recurrent pterygium | 6 months
  severity score of impending recurrent pterygium included 3 factors; redness, thickness of fibrovascular tissue, and size of fibrovascular tissue at 3 mm from limbus, which are classified into 3 grades in each factor.
time to recurrent of pterygium | 6 months
  time from enrolled participants until they developed true recurrent pterygium
rate of steroid induced ocular hypertension | 6 months
  number of participants in each group who had intraocular pressure > 21 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Wannisa Suphachearabhan, MD, Principal Investigator — Srinakharinwirot University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mahar PS, Manzar N. Pterygium recurrence related to its size and corneal involvement. J Coll Physicians Surg Pak. 2013 Feb;23(2):120-3. PMID 23374515
- [Result] Sherwin JC, Hewitt AW, Kearns LS, Griffiths LR, Mackey DA, Coroneo MT. The association between pterygium and conjunctival ultraviolet autofluorescence: the Norfolk Island Eye Study. Acta Ophthalmol. 2013 Jun;91(4):363-70. doi: 10.1111/j.1755-3768.2011.02314.x. Epub 2011 Dec 16. PMID 22176664
- [Result] Yaisawang S, Piyapattanakorn P. Role of post-operative topical corticosteroids in recurrence rate after pterygium excision with conjunctival autograft. J Med Assoc Thai. 2003 Jun;86 Suppl 2:S215-23. PMID 12929992
- [Result] Hirst LW. The treatment of pterygium. Surv Ophthalmol. 2003 Mar-Apr;48(2):145-80. doi: 10.1016/s0039-6257(02)00463-0. PMID 12686302
- [Result] Kucukerdonmez C, Akova YA, Altinors DD. Comparison of conjunctival autograft with amniotic membrane transplantation for pterygium surgery: surgical and cosmetic outcome. Cornea. 2007 May;26(4):407-13. doi: 10.1097/ICO.0b013e318033b3d4. PMID 17457187
- [Result] Pikkel J, Porges Y, Ophir A. Halting pterygium recurrence by postoperative 5-fluorouracil. Cornea. 2001 Mar;20(2):168-71. doi: 10.1097/00003226-200103000-00011. PMID 11248822
- [Result] Anguria P, Ntuli S, Carmichael T. Young patient's age determines pterygium recurrence after surgery. Afr Health Sci. 2014 Mar;14(1):72-6. doi: 10.4314/ahs.v14i1.11. PMID 26060460
- [Result] Han SB, Jeon HS, Kim M, Lee SJ, Yang HK, Hwang JM, Kim KG, Hyon JY, Wee WR. Risk Factors for Recurrence After Pterygium Surgery: An Image Analysis Study. Cornea. 2016 Aug;35(8):1097-103. doi: 10.1097/ICO.0000000000000853. PMID 27100658
- [Result] Olusanya BA, Ogun OA, Bekibele CO, Ashaye AO, Baiyeroju AM, Fasina O, Ogundipe AO, Ibrahim AO. Risk factors for pterygium recurrence after surgical excision with combined conjunctival autograft (CAG) and intraoperative antimetabolite use. Afr J Med Med Sci. 2014 Mar;43(1):35-40. PMID 25335376
- [Result] Nuzzi R, Tridico F. How to minimize pterygium recurrence rates: clinical perspectives. Clin Ophthalmol. 2018 Nov 19;12:2347-2362. doi: 10.2147/OPTH.S186543. eCollection 2018. PMID 30538417
- [Result] Kim KW, Kim JC. Current approaches and future directions in the management of pterygium. Int J Ophthalmol. 2018 May 18;11(5):709-711. doi: 10.18240/ijo.2018.05.01. eCollection 2018. PMID 29862166
- [Result] Prabhasawat P, Tesavibul N, Leelapatranura K, Phonjan T. Efficacy of subconjunctival 5-fluorouracil and triamcinolone injection in impending recurrent pterygium. Ophthalmology. 2006 Jul;113(7):1102-9. doi: 10.1016/j.ophtha.2006.02.026. Epub 2006 May 26. PMID 16730066
- [Result] Makornwattana M, Suphachearaphan W. Incidence of steroid induced-ocular hypertension in postoperative pterygium excision. J Med Assoc Thai. 2015 Mar;98 Suppl 2:S151-7. PMID 26211117
- [Result] Bodor N, Buchwald P. Soft drug design: general principles and recent applications. Med Res Rev. 2000 Jan;20(1):58-101. doi: 10.1002/(sici)1098-1128(200001)20:13.0.co;2-x. PMID 10608921
- [Result] Comstock TL, Sheppard JD. Loteprednol etabonate for inflammatory conditions of the anterior segment of the eye: twenty years of clinical experience with a retrometabolically designed corticosteroid. Expert Opin Pharmacother. 2018 Mar;19(4):337-353. doi: 10.1080/14656566.2018.1439920. Epub 2018 Mar 7. PMID 29430976
- [Result] Sheppard JD, Comstock TL, Cavet ME. Impact of the Topical Ophthalmic Corticosteroid Loteprednol Etabonate on Intraocular Pressure. Adv Ther. 2016 Apr;33(4):532-52. doi: 10.1007/s12325-016-0315-8. Epub 2016 Mar 17. PMID 26984315